CLINICAL TRIAL: NCT01391338
Title: A Phase II, Randomized, Double-blind, Placebo-controlled, Parallel Group, Adaptive, Combined Proof of Concept and Dose-Finding Study to Investigate Efficacy, Safety, Pharmacodynamics and Pharmacokinetics of ASP3652 in the Treatment of CP/CPPS
Brief Title: A Clinical Study to Investigate the Efficacy, Safety and Pharmacokinetics of ASP3652 in Patients With Chronic Abacterial Prostatitis / Chronic Pelvic Pain Syndrome (CP/CPPS)
Acronym: AZURE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3652-CL-0019; 2010-023775-25 (EudraCT Number)
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Abacterial Prostatitis; Chronic Pelvic Pain Syndrome
Keywords: Prostatitis; Chronic; Pelvic Pain; NIH-CPSI; Pain domain score in NIH-CPSI
MeSH Terms: conditions — Prostatitis; Bronchiolitis Obliterans Syndrome; Pelvic Pain | interventions — ASP3652

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Lowest dose ASP3652 twice daily (Experimental)
  Interventions: Drug: ASP3652
- Low dose ASP3652 twice daily (Experimental)
  Interventions: Drug: ASP3652
- Medium dose ASP3652 twice daily (Experimental)
  Interventions: Drug: ASP3652
- High dose ASP3652 once daily (Experimental)
  Interventions: Drug: ASP3652
- High dose ASP3652 twice daily (Experimental)
  Interventions: Drug: ASP3652
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP3652 — Oral
  Arms: High dose ASP3652 once daily; High dose ASP3652 twice daily; Low dose ASP3652 twice daily; Lowest dose ASP3652 twice daily; Medium dose ASP3652 twice daily
Drug: Placebo — Oral
  Arms: Placebo

SUMMARY:
In this study several doses of ASP3652, given orally for 12 weeks, will be compared with placebo in the treatment of patients with Chronic abacterial Prostatitis / Chronic Pelvic Pain Syndrome.

DETAILED DESCRIPTION:
This study will investigate the efficacy of ASP3652 in the treatment of patients with Chronic abacterial Prostatitis / Chronic Pelvic Pain Syndrome (CP/CPPS). In comparison with placebo, ASP3652 will be given in different dosages orally for 12 weeks. The aims are to investigate efficacy of ASP3652 in CP/CPPS, to assess the optimal dose of ASP3652, to investigate safety and tolerability and to investigate pharmacokinetics and pharmacodynamics of ASP3652 in patients with CP/CPPS in and out-patients setting.

ELIGIBILITY:
Inclusion Criteria:

* Is diagnosed with CP/CPPS with symptoms for at least 3 months over the last 6 months
* Has a NIH-CPSI total score of at least 15
* A score of at least 4 on question 4 (pain) in the NIH-CPSI
* Reports pain on palpation of the prostate or the perineum/genital area
* Answers "yes" to at least 1 out of 6 items in question 1 and 2 of the NIH-CPSI
* Is willing to comply with study requirements such as completing the micturition and symptoms diary and attend all study visits

Exclusion Criteria:

* Isolated unilateral testicular, penile or scrotal pain as a solitary symptom of pelvic pain
* Urinary Tract Infection (UTI) or prostate infection found at screening using the pre- and post massage test or in the last 3 months prior to screening
* Any prior prostate and or bladder intervention within 3 months prior to screening
* Lower urinary tract malignancy (suspected), such as positive (micro) hematuria in urine sediment or Prostate Specific Antigen (PSA) >4 ng/mL
* Symptomatic urethral stricture or symptomatic bladder or urethral calculi, severe bladder outlet obstruction, overactive bladder with incontinence or Post Void Residual volume, greater than 150 mL
* Clinically significant abnormalities on transabdominal ultrasound of bladder and prostate or neurological disease or defect affecting bladder function
* Currently active sexually transmittable disease
* Substance abuse or any use of delta-9-tetrahydrocannabinol (THC) as assessed by a positive urine test for THC at screening
* Major depression, i.e. a Center for Epidemiological Studies Depression Scale score of 27 or more
* Any clinically relevant concomitant disease (past or present) which would, in the opinion of the investigator, put the subject at risk or mask measures of efficacy
* Use of steroids, immunomodulators, anticonvulsants, cytochrome P4502C8 inhibitors, cannabis/THC based medication, opioid analgetics or antiviral/antimicrobial/antifungal agents during the last 4 weeks before screening
* Initiation, discontinuation, or variation in the dose of antidepressants, alpha-blockers, 5-alpha reductase inhibitors, antimuscarinics, benzodiazepines, skeletal muscle relaxants, non-steroidal antiinflammatory drugs, non-opioid analgetics and herbal therapies during the last 4 weeks before screening. Subjects should continue these medications at that same stable dose throughout the study
* Clinically relevant abnormal urine or blood safety laboratory values or active hepatic and/or biliary disease (AST or ALT should not be >3 times the upper limit of normal, total bilirubin should not be >2 times the upper limit of normal)
* Participated in any clinical study or has been treated with any investigational drug or device within 30 days prior to screening, or the period stipulated by local regulations, whichever is longer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the National Institutes of Health-Chronic Prostatitis Symptom Index (NIH-CPSI), total score at 12 weeks | Baseline and 12 weeks

SECONDARY OUTCOMES:
Change from baseline in the NIH-CPSI pain domain score at week 12 | Baseline and 12 weeks
Change from baseline in NIH-CPSI total score at 4 and 8 weeks and at 2 weeks follow-up after treatment | Baseline, 4 weeks, 8 weeks and 2 weeks follow-up post treatment
Change from baseline in NIH-CPSI pain domain at week 4 and 8 and at 2 weeks follow-up after treatment | Baseline, 4 weeks, 8 weeks 2 weeks follow-up post treatment
Change from baseline in NIH-CPSI urinary symptoms domain at week 4, 8 and 12 and at 2 weeks follow-up after treatment | Baseline, 4 weeks, 8 weeks and 12 weeks treatment and weeks 2 weeks follow-up post treatment
Change from baseline in NIH-CPSI Quality of Life impact domain at week 4, 8 and 12 and at 2 weeks follow-up after treatment | Baseline, 4 weeks, 8 weeks and 12 weeks treatment and weeks 2 weeks follow-up post treatment
Global Response Assessment at week 4, 8 and 12 and at 2 weeks follow-up post treatment | Baseline, 4 weeks, 8 weeks and 12 weeks treatment and at 2 weeks follow-up post treatment
The proportion of Clinical Responders | 12 weeks
  Composite of two definitions are used: subjects who showed at least 4 points decrease in NIH-CPSI total score at 12 weeks compared to baseline and subjects who showed at least 6 points decrease in NIH-CPSI total score at 12 weeks
Genitourinary pain index (GUPI) total score, sub domain and responders, at week 12 | 12 weeks
  Responder defined as 7 points or more decrease from baseline
Mean daily CPSI-24hour total score at baseline and at 4, 8 and 12 weeks and 2 weeks follow-up post treatment | Baseline, 4 weeks, 8 weeks and 12 weeks and 2 weeks follow-up post treatment
Mean daily pain for the 7 days period prior to attending study visits at baseline and at 4, 8 and 12 weeks and 2 weeks follow-up post treatment | Baseline, 4 weeks, 8 weeks and 12 weeks and 2 weeks follow-up post treatment
Short form McGill pain questionnaire: sensory, affective and total score, VAS, present pain intensity at baseline and at 12 weeks | Baseline and 12 weeks
Voiding: mean number of micturitions per 24 hours and per night, mean number of urgency episodes per 24 hours and mean level of urgency per micturition | Baseline, 4 weeks and 12 weeks treatment
  Based on daily urinary symptom diary for 3 consecutive days in the weeks prior to the visits at baseline, 4 and 12 weeks treatment
International Prostate Symptom Score at screening and at 12 weeks | Screening and 12 weeks
European Quality of Life questionnaire in 5 dimensions (EQ-5D) at baseline and at 12 weeks | Baseline and 12 weeks
Male sexual health questionnaire at baseline and at 12 weeks | Baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Executive Director Global Medical Science, Study Director — Astellas Pharma Europe B.V.; Coordination Investigator, Principal Investigator — Clinic for Urology, Pediatric Urology and Andrology, Germany
Locations (49):
- Czechia (12):
  - Site: 3105 - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Site: 3106 - Urologicke oddeleniUsti nad Labem, Kolín
  - Site: 3109- Hospital Kromeriz, Kroměříž
  - Site: 3107 - Urologie, Nový Jičín
  - Site: 3103 - Fakultni nemocnice Olomouc, Olomouc
  - Site: 3111 - Urology center, Pilsen
  - Site: 3112 - Urosante, Prague
  - Site: 3102 - Androgeos, Prague
  - Site: 3110 - Urologicka ordinace, Sternberk
  - Site: 3104 - Uherskohradistska nemocnice a.s., Uherské Hradiště
  - Site: 3101- Krajska zdravotni, a.s. - Masarykova nemocnice v Usti nad Labem, o.z., Ústí nad Labem
  - Site: 3113 - Urologicka ambulance, Žatec
- Germany (15):
  - Site: 3212 - Urologische Praxis, Berlin
  - Site: 3214 - Charité Campus Benjamin Franklin, Berlin
  - Site: 3208 - Private Praxis Urologie Borken, Borken
  - Site: 3202 - Urologische Praxis, Buchholz
  - Site: 3201 - Universitats klinikum Giessen und Marburg, Giessen
  - Site: 3203 - Urologische Praxis, Hamburg
  - Site: 3211 - Urologische Gemeinschaftspraxis, Herzogenaurach
  - Site: 3205 - Gesundheitszentrum Holzminden, Holzminden
  - Site: 3213 - Urologische Praxis, Kempen
  - Site: 3206 - Private Praxis, Leipzig
  - Site: 3210 - Private Praxis, Marburg
  - Site: 3207 - Private Praxis, Markkleeberg
  - Site: 3204 - Akademisches Lehrkrankenhaus, Neunkirchen
  - Site: 3215 - Urologische Praxis, Reutlingen
  - Site: 3209 - Private Praxis, Sangerhausen
- Latvia (4):
  - Site: 3302 - Jelgava Outpatient Clinic, Jelgava
  - Site: 3301 - Litavniece Urologist Private Practice, Liepāja
  - Site: 3303 - P. Stradins Clinical University Hospital, Riga
  - Site: 3304 - Nord Kurzeme Regional Hospital, Ventspils
- Lithuania (4):
  - Site: 3404 - Motina ir vaikas clinic, Kaunas
  - Site: 3402 - Vilnius Univeristy Hospital "Santariskiu Klinikos" Urology Centre, Vilnius
  - Site: 3401 - Clinics "Privatus gydytojas", Vilnius
  - Site: 3403 - Public Institution Vilnius City University Hospital, Vilnius
- Poland (11):
  - Site: 3503 - Urovita Sp.z.o.o. NZOZ Szpital Slaskie Centrum Urologii, Chorzów
  - Site: 3504 - Centrum Medyczne Szpital Sw Rodziny Sp z o.o., Lodz
  - Site: 3509 - NZOZ Nasz Lekarz, Praktyka Grupowa Lekarzy Rodzinnych z Przychodnia Specjalistyczna, Lotum
  - Site: 3510 - Heureka Hanna Szalecka, Piaseczno
  - Site: 3501 - Indywidualna Specjalistyczna Praktyka Lekarska, Poznan
  - Site: 3511 - Urologica Praktyka Lekarska Adam Marcheluk, Siedlce
  - Site: 3508 - NZOZ Centrum Medyczna Wola, Warsaw
  - Site: 3507 - Szpital Kliniczny Dzieciatka Jezus Centrum Leczenia Obrazen, Warsaw
  - Site: 3502 - Wojewodzki Szpital Specjalistyczny we Wroclawiu, Wroclaw
  - Site: 3505 - EMC Instytut Medyczny SA, Wroclaw
  - Site: 3506 - Specjalistyczna Praktyka Lekarska Gabinet Urologiczny, Wroclaw
- Spain (3):
  - Site: 3701 - Hospital Moises Broggi de Sant Joa, Barcelona
  - Site: 3703 - Fundació Puigvert, Barcelona
  - Site: 3702 - Hospital del Henares, Coslada

REFERENCES:
- [Derived] Martina R, Houbiers J, Melis J, van Till O. A combined proof of concept and dose finding study with multiple endpoints: A Bayesian adaptive design in chronic prostatitis/chronic pelvic pain syndrome. Biom J. 2019 May;61(3):476-487. doi: 10.1002/bimj.201700210. Epub 2018 Sep 3. PMID 30178528